CLINICAL TRIAL: NCT03801109
Title: Study of the Effectiveness of Transcranial Magnetic Stimulation and the Hyperbaric Chamber in Women With Fibromyalgia. Randomized Clinical Trial.
Brief Title: Transcranial Magnetic Stimulation and Hyperbaric Chamber for Women Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: H1548771544856
Record Dates: First submitted 2018-11-14; First posted 2019-01-11 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2019-12

CONDITIONS: Fibromyalgia
Keywords: transcranial magnetic stimulation; hyperbaric chamber; pain; endorphins
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hyperbaric group (Experimental)
  Interventions: Other: Hyperbaric group
- Magnetic group (Experimental)
  Interventions: Other: Magnetic group
- Physical group (Active Comparator)
  Interventions: Other: Physical group; Other: Baseline group
- Baseline group (No Intervention)

INTERVENTIONS:
Other: Hyperbaric group — Participants in this group performed 5 sessions per week for 8 weeks (40 sessions in total) . The time of each session is 90 minutes and the chamber pressure is 1.4 ATA with a 100% oxygen mask.
  Arms: Hyperbaric group
Other: Magnetic group — There will be 5 sessions per week for 2 consecutive weeks (10 sessions in total), stimulating the left motor cortex at high frequencies, 10 Hz, for 30 minutes.
  Arms: Magnetic group
Other: Physical group — A protocol of low-impact physical exercise will be performed twice a week for 8 weeks, with a total of 16 sessions.
  Arms: Physical group
Other: Baseline group — This group will be the control group that did not take any action, perform the activities of daily life
  Arms: Physical group

SUMMARY:
Fibromyalgia syndrome (FMS) is a multisystem disease, characterized by generalized chronic musculoskeletal pain. In addition, there is a lot of care for fatigue, sleep disorders, morning stiffness, cognitive disorders, depression, anxiety and stress. Other common symptoms are back pain, headaches, irritable bowel, balance problems and deterioration of physical function in general. Patients with fibromyalgia (FM) often show pain at specific points that are known as "tender spots or tender spots, with an increased sensitivity to painful stimuli" (hyperalgesia) and a decreased pain threshold (allodynia). which can be evidenced in the physical examination and in the absence of anomalies that justify in the biological or image tests. These pain points to pressure, based on the most specific and specific criteria for the diagnosis of the disease, traditionally based on the criteria of the American College of Rheumatology (ACR), according to which, should be presented so minus 11 out of 18 painful points to confirm it. Although the etiology remains unknown and unclear, its appearance is attributed to a problem of central sensitization, that is, changes in central processing, which causes an alteration of the mechanisms that regulate the sensation of pain, with amplification of nociceptive input . and perpetuation of painful stimuli. Fibromyalgia is becoming a common syndrome in the countries of Western Europe, with a prevalence in the general population that ranges between 1-3%, and specifically in Spain, around 2.4%. In addition, it has a higher incidence in women than men (73-95%), predominantly affecting women between the ages of 40-50 years. About 3% of women with fibromyalgia are at an age when menopause occurs, so not only do they experience the symptoms of both states but they even exacerbate the syndrome with each other. On the other hand, and in relation to its chronicity, the care of this type of patients involves large costs for society with a significant consumption of health resources in the field of primary care, as well as the costs of work absenteeism. For these reasons, it is considered an important problem with a great impact on the health system, and therefore more and more studies are being developed with the aim of better understanding the pathophysiology of this disease. The therapeutic approach includes low cost and easy access measures, such as physical exercise (EF) programs to improve the symptoms of FM. Physical exercise has positive effects directly on pain, joint and muscle stiffness, generalized sensitivity and fatigue, among others, and secondarily on cognitive disorders. Thus, the vast majority of studies focus on low-impact aerobic exercise, performed between 60% and 70% of the maximum heart rate two to three times a week. However, to date, there is no study that compares the effectiveness of physical exercise with other innovative therapeutic actions, such as transcranial magnetic stimulation (TMS), the hyperbaric chamber (HBOT), in parameters related to pain and quality of life. the life of patients with fibromyalgia. The general objective is the effectiveness of transcranial magnetic stimulation and the hyperbaric chamber in women with fibromyalgia. As specific objectives we propose:

To assess the effect of HBOT, TMS and EF on quality of life in women with fibromyalgia.

* Object the effect of HBOT, TMS and EF in cortical functioning.
* Evaluate the effect of HBOT, TMS and EF on fatigue.
* Evaluate the effect of HBOT, TMS and EF on psychological aspects, such as depression and anxiety.
* Evaluate the effect of HBOT, TMS and EF on the perception of pain and the number of painful points.
* Evaluate the effect of HBOT, TMS and EF on the quality of sleep.
* Evaluate the effect of HBOT, TMS and EF on the quality of life.
* Evaluate the effect of HBOT, TMS and EF on the pain constructs.
* Determine the effect of HBOT, TMS and EF on plasma endorphin levels.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Fibromyalgia according to the criteria of the American College of Rheumatology of 1990.
* Having taken pharmacological treatment for more than three months without clinical improvement.
* Have the capacity to sign the informed consent form in accordance.
* Not having previously received treatment with a hyperbaric chamber or transcranial magnetic stimulation.
* Absence of other pathologies associated with the locomotor system at an advanced stage that makes physical activity impossible (arthritis, osteoarthritis, uric acid).

Exclusion Criteria:

* Pregnancy or lactation period.
* Epilepsy, drugs that lower the convulsive threshold, history of intense headaches, e endocranial and auditory elements, pathology related to the nervous system, either central or peripheral, not associated with fibromyalgia, endocranial hypertension.
* Hospital hypertension not controlled, heart and / or respiratory failure, cardiac pacemaker, pneumothorax.
* Claustrofobia and / or psychiatric pathologies; schizophrenia, bipolar disorder, psychosis.
* Patients with problems of alcohol addiction, psychoactive drugs or narcotics.
* Patients presenting neoplasia.
* Surgical interventions of less than 4 months.
* Tympanic perforations.
* Cardiac slides.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Changes in pain intensity | Hyperbaric, Physical and Baseline groups: change from baseline in the intensity of pain at 8 weeks. Magnetic group: change from baseline in the intensity of pain at 3 weeks.
  Analog visual scale

SECONDARY OUTCOMES:
Rating of pain | Hyperbaric, Physical and Baseline groups: baseline and 8 weeks. Magnetic group: baseline and 3 weeks
  The McGill Pain Questionnaire can be used to evaluate a person experiencing significant pain. Interpretation : 0 minimum pain score and 78 maximum pain score. The higher the pain score the greater the pain.
Pain catastrophizing | Hyperbaric, Physical and Baseline groups: baseline and 8 weeks. Magnetic group: baseline and 3 weeks
  it will be measurde by pain catastrophizing scale. It is a Self-administered scale on a 5-point Likert scale ranging from 0 (never) to 4 (always), which are distributed in 3 subscales: rumination (refers to a state or feeling of constant worry and the inability to inhibit thoughts related to pain), despair (manifested when hope has been lost for achieving something, or because it disappears or because it gives off some physical and / or psychological aspect that is detrimental to health) and magnification (refers to the exaggeration of unpleasant situations of pain and expectations of negative consequences). Higher scores indicate higher levels of catastrophism.
Acceptance of pain | Hyperbaric, Physical and Baseline groups: baseline and 8 weeks. Magnetic group: baseline and 3 weeks
  The Chronic Pain Acceptance Questionnaire (CPAQ) is a 20-item inventory designed to measure acceptance of pain. here are two principle factors measured by this questionnaire: activities engagement and pain willingness. All items are rated on a 0 (never true) to 6 (always true) scale. The maximum possible total score is 120, with a higher score indicating better acceptance
Pain self perception | Hyperbaric, Physical and Baseline groups: baseline and 8 weeks. Magnetic group: baseline and 3 weeks
  The Pain Self-Perception Scale (PSPS) is a 24-item questionnaire used to assess mental defeat in chronic pain patients. espondents are asked to indicate to what extent each of the 24 statements applied to their experience "during a recent episode of intense pain". These statements are to be rated on a 5-point scale (0 = "Not at all/Never," 1 = "Very little," 2 = "Moderately," 3 = "Strongly," 4 = "Very strongly"), generating a total score ranging from 0 to 96. a higher score indicating worst self perception
Psychological inflexibility | Hyperbaric, Physical and Baseline groups: baseline and 8 weeks. Magnetic group: baseline and 3 weeks
  The scale that will be used is the Psychological Inflexibility in Pain Scale. It is a 12-item scale designed to measure psychological inflexibility in pain patients.The items consisted of different statements that were considered to be related to chronic pain, psychological inflexibility, suffering and disability All of the items were rated on a 7-point Likert-type scale that ranged from "1=never true" to "7=always true", with higher scores indicating more psychological inflexibility.
Number of painful points | Hyperbaric, Physical and Baseline groups: baseline and 8 weeks. Magnetic group: baseline and 3 weeks
  The sensitivity of the 18 trigger points originally defined in the diagnosis of Fibromyalgia will be studied by means of an FPX 25 algometer (Wagner Instruments, Greenwich, USA) that records the pain threshold experienced
Quality of life: perceived well-being | Hyperbaric, Physical and Baseline groups: baseline and 8 weeks. Magnetic group: baseline and 3 weeks
  SF-12 Satisfacción with life scale
Quality of sleep | Hyperbaric, Physical and Baseline groups: baseline and 8 weeks. Magnetic group: baseline and 3 weeks
  Epworth Sleepiness Scale: the instrument asks the researched subject, about the frequency (or probability) of falling asleep on a scale of increase that from 0 to 3, for eight different daily situations, that most people can be involved, in your daily life, although not necessarily every day.2 The score of the 8 situations is added to obtain a total number. A result between 0 and 9 is considered normal; while one between 10 and 24 indicates that the patient should be referred to a specialist.
Level of depression | Hyperbaric, Physical and Baseline groups: baseline and 8 weeks. Magnetic group: baseline and 3 weeks
  The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. items are rated on a 4-point scale ranging from 0 to 3 based on severity of each item. The maximum total score is 63. Higher punctuations meaning, Higher scores indicate that the degree of depression is more severe
Level of stress | Hyperbaric, Physical and Baseline groups: baseline and 8 weeks. Magnetic group: baseline and 3 weeks
  To assess the state of stress the scale will be used the perceived srtress scale. This scale is a self-report instrument that evaluates the level of stress perceived during the last month, consists of 14 items with a response format of a scale of five points (0 = never, 1 = almost never, 2 = from time to time). when, 3 = often, 4 = very often). The total score of the PSS is obtained by inverting the scores of items 4, 5, 6, 7, 9, 10 and 13 (in the following sense: 0 = 4, 1 = 3, 2 = 2, 3 = 1 and 4 = 0) and then adding the 14 items. The direct score obtained indicates that a higher score corresponds to a higher level of perceived stress.
Level of anxiety | Hyperbaric, Physical and Baseline groups: baseline and 8 weeks. Magnetic group: baseline and 3 weeks
  To assess the state of stress the scale will be used the Hospital Anxiety and Depression Scale, it is a self-applied questionnaire with 14 items, on a Likert scale of 0-3. Higher score, greater anxiety and depression.
Evoked motor potential | Hyperbaric, Physical and Baseline groups: baseline and 8 weeks. Magnetic group: baseline and 3 weeks
  The evoked motor potential will be recorded in each subject through the Neuro-MEP-Micro EMG, with the Neuro-MEO.NETomega.3.7.3.7 software. and surface electrodes placed in the musculature of the first dorsal interosseous. In addition, after acquiring the resting motor threshold of each subject, we have obtained the motor power evoked at 120 and 140%, to calculate the ratio of the amplitude of the potential.
Motor threshold | Hyperbaric, Physical and Baseline groups: baseline and 8 weeks. Magnetic group: baseline and 3 weeks
  The resting motor threshold is defined as the minimum signal strength that must be provided to have an evoked motor potential of at least 50 microvolts in 50% of the tests. In our study we used the software TMS_MTAT_2.0.1 to calculate by means of an algorithm which is the minimum intensity of each subject, in the first dorsal interosseous of the right hand. To obtain it, a stimulation of a simple puslo will be carried out using the neuro-MS / D magnetic stimulator. Placed in the motor cortex M1, at 45º orientation with respect to the midline.
Plasma pain biomarkers. | Hyperbaric, Physical and Baseline groups: baseline and 8 weeks. Magnetic group: baseline and 3 weeks
  Beta-endorphin concentrations (pg/mL) will be measured by Human β-EP(Beta-Endorphin) ELISA Kit. The concentration ofHumanβ-EPin the samples is then determined by comparing the optical density (OD) of the samples to the standard curve

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Izquierdo Alventosa, PT, Principal Investigator — University of Valencia
Locations (1):
- Fundación Fivan, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Izquierdo-Alventosa R, Ingles M, Cortes-Amador S, Munoz-Gomez E, Molla-Casanova S, Gimeno-Mallench L, Chrivella-Garrido J, Serra-Ano P. Effects of a low-pressure hyperbaric oxygen therapy on psychological constructs related to pain and quality of life in women with fibromyalgia: A randomized clinical trial. Med Clin (Barc). 2024 Jun 14;162(11):516-522. doi: 10.1016/j.medcli.2023.12.016. Epub 2024 Feb 20. English, Spanish. PMID 38383268
- [Derived] Izquierdo-Alventosa R, Ingles M, Cortes-Amador S, Gimeno-Mallench L, Sempere-Rubio N, Serra-Ano P. Effectiveness of High-Frequency Transcranial Magnetic Stimulation and Physical Exercise in Women With Fibromyalgia: A Randomized Controlled Trial. Phys Ther. 2021 Oct 1;101(10):pzab159. doi: 10.1093/ptj/pzab159. PMID 34216139
- [Derived] Izquierdo-Alventosa R, Ingles M, Cortes-Amador S, Gimeno-Mallench L, Sempere-Rubio N, Chirivella J, Serra-Ano P. Comparative study of the effectiveness of a low-pressure hyperbaric oxygen treatment and physical exercise in women with fibromyalgia: randomized clinical trial. Ther Adv Musculoskelet Dis. 2020 Jun 24;12:1759720X20930493. doi: 10.1177/1759720X20930493. eCollection 2020. PMID 32636943